CLINICAL TRIAL: NCT02759237
Title: The Medtronic Transcatheter Aortic Valve Implant System (CoreValve System Family) Post Marketing Surveillance (PMS) (CoreValve India PMS)
Acronym: CoreValveIndia
Status: Terminated | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Version 1.0 17 February 2016; REF/2016/04/011112 (Other: Clinical Trials Registry - India)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Symptomatic Aortic Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient Group: Patients identified for treatment of symptomatic aortic sten
  Interventions: Device: CoreValve System Family

INTERVENTIONS:
Device: CoreValve System Family — Bioprosthesis: Transcatheter Aortic Valve Implant (TAV - Heart Valve) -Different Models/Sizes of CoreValve/CoreValve Evolut R.
  Delivery Catheter System: ACCUTRAK & EnVeo R - Used to facilitate the placement of the bioprosthesis within the annulus.
  Loading System: Compression Loading System & EnVeo R Loading System - Used to load the TAV onto the delivery system
  Other Names: Medtronic Transcatheter Aortic Valve Implant System (CoreValve System Family)

SUMMARY:
The Medtronic Transcatheter Aortic Valve Implant System (CoreValve System Family) has been demonstrated to be safe and effective for high through extreme risk patients with symptomatic severe native aortic stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure. Per DCGI systematic post marketing surveillance requirement, the purpose of this PMS plan is to provide local post marketing surveillance data regarding the safety of Medtronic CoreValve System Family

DETAILED DESCRIPTION:
The objective of this PMS will be to monitor and gather data on the safety of The Medtronic Transcatheter Aortic Valve Implant System (CoreValve System Family) in the approved intended use.

The main focus of this PMS will be to generate additional information and report on all major adverse events up to 30 days from the day of implant procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic heart disease due to severe native calcific aortic stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure and with anatomy appropriate for the 23, 26, 29 or 31 mm valve system who are judged by a heart team, including a cardiac surgeon, to be at high or greater risk for open surgical therapy.
* Indications and contraindications are provided in the product Instructions for Use.
* Subject is scheduled to receive transcatheter aortic valve
* Subject is 18 years of age or older
* The patient or his/her Legally Authorized Representative (LAR) has been informed about the nature of the PMS and the Informed consent for both Audio Visual (AV) recording and for study participation has been obtained prior to performing any study-related procedures from the subject or Legally Authorized Representative, as per applicable local requirements in India

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified for treatment of symptomatic aortic stenosis (AS), necessitating The Medtronic Transcatheter Aortic Valve Implant System (CoreValve System Family) as part of standard of care, in accordance with the product label indications (Instructions for Use), contraindications, and warnings
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Safety outcomes: all major adverse events | 30 days post procedure
  This is a surveillance plan designed to collect and report safety outcomes; hence there are no additional clinical endpoints identified. The main focus of this PMS will be to generate additional information and report on all major adverse events up to 30 days from the day of implant procedure.
MACCE | 30 day post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Acute kidney Injury | 30 day post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Cardiac tamponade | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Prosthetic valve dysfunction - including moderate or severe aortic regurgitation | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Cardiogenic shock | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Prosthetic valve endocarditis | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Life-threatening, disabling or major bleeding | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Major vascular complication | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Cardiac perforation | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Valve malpositioning | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure
Thrombosis and coronary occlusion | 30 days post procedure
  Safety endpoints will be reported as Kaplan-Meier rates which are probabilities of having an event at 30 days post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Eternal Heart Care Centre, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: No